CLINICAL TRIAL: NCT01899677
Title: The Efficacy of Symbiotic Preparation on Cytokines Which Act on Necrotising Enterocolitis Pathogenesis in Very Low Birth Weight Infants
Brief Title: The Efficacy of Symbiotic on Cytokines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ozge Serce, specialist in neonatology, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14893
Record Dates: First submitted 2013-07-01; First posted 2013-07-15 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Necrotising Enterocolitis
Keywords: Symbiotic,cytokines, necrotising enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- symbiotic (Experimental): symbiotic preparation 1/2 sachet twice daily during 30 days
  Interventions: Drug: symbiotic
- distilled water (Placebo Comparator): 2 x 0.5 cc distilled water will be given during 30 days
  Interventions: Other: distilled water

INTERVENTIONS:
Other: distilled water — 0.5 cc distilled water twice daily will be added to the breast milk or formula during 30 days
  Arms: distilled water
Drug: symbiotic — Symbiotic 1/2 sachet twice daily will be added to the breast milk or formula during 30 days
  Other Names: Probiotic ATP
  Arms: symbiotic

SUMMARY:
The aim of this prospective double blinded randomised study is to investigate the efficacy of symbiotic preparation which contains lactobacillus casei, L. rhamnosus, L. plantarum, Bifidobacterium lactis, fructo and galactooligosaccharide on cytokines as interferon-gama acting on Th1 pathway, interleukin -5 acting on Th2, interleukin -10 acting on T regulatory pathway, and interleukin -17 acting on Th-17 pathway that were related with necrotizing enterocolitis pathogenesis in very low birth weight neonates.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Neonates who born 26- 32 gestational week and 750-1500 gram birth weights
2. Neonates who tolerated minimal enteral feeding within postnatal first week

Exclusion criteria:

1. PROM> 24 hours and/or chorioamnionitis
2. Mechanic ventilation supply more than 7 days
3. Culture proven sepsis
4. Major congenital anomaly
5. Patients undergoing surgery

Intervention:

The allocations will contain in opaque, sequentially numbered sealed envelopes. The study group will receive symbiotic preparation (Probiotic ATP, Nobel, 1/2 sachet twice daily); whereas the control group will receive placebo (distilled water; 1 ml per dose twice daily) which will be added to breast milk or formula starting with the first feed.0.5 cc blood sampling will be taken from patients within postnatal 48 hours, 14+2.days, 28+2.days. This samples will turn by cold centrifugation and store at -20 °C temperature. The cytokines will be analysed by ELISA multiplex method.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates born 26- 32 gestational weeks and 750-1500 gram birth weights
2. Neonates who tolerated minimal enteral feeding during first week of life

Exclusion Criteria:

1. PROM> 24 hour and/or chorioamnionitis
2. Mechanical ventilation supply more than 7 days
3. Culture proven sepsis
4. Major congenital anomaly
5. Neonates undergoing surgery

Ages: 1 Hour to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fahri Ovali, Study Director — Zeynep Kamil Maternity and Childen Education and Training Hospital; Ozge Serce, Principal Investigator — Zeynep Kamil Maternity and Childen Education and Training Hospital; Tugba Gursoy, MD, Study Chair — Zeynep Kamil Maternity and Children Education and Training Hospital
Locations (1):
- Zeynep Kamil Maternity and Child Health Hospital, Istanbul, Umraniye, Turkey (Türkiye)

REFERENCES:
- [Background] Ng SC, Hart AL, Kamm MA, Stagg AJ, Knight SC. Mechanisms of action of probiotics: recent advances. Inflamm Bowel Dis. 2009 Feb;15(2):300-10. doi: 10.1002/ibd.20602. PMID 18626975

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symbiotic | Distilled Water
Started | 35 | 35
Completed | 25 | 28
Not Completed | 10 | 7

BASELINE CHARACTERISTICS:
Population: Very low birth weight neonates
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbiotic | Distilled Water | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 28 | 53
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 12 | 18 | 30
birth weight [Mean (Standard Deviation); unit: grams] | 1266 (228) | 1230 (262) | 1245 (247)

OUTCOME MEASURES:

1. Primary Outcome: Interleukin 5 Serum Cytokine Level on 0+2 Day
Time Frame: 0+2 day
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 4 [2.5 to 5.5] | 4 [2 to 4]
Statistical Analysis 1: Comparison: Symbiotic vs Distilled Water; Mann Whitney U test was used to compare cytokine levels between groups; Test type: Superiority or Other; p = 0.32, Mann whitney U

2. Primary Outcome: Interleukin 5 Levels on 14+/-2 Day
Time Frame: 14+/-2 day
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 4 [2.5 to 7.5] | 4 [2.2 to 11.2]
Statistical Analysis 1: Comparison: Symbiotic vs Distilled Water; Test type: Superiority or Other; p = 0.73, Mann whitney U

3. Primary Outcome: Interleukin 5 Levels at 28+/-2 Day
Time Frame: 28+/-2 day
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 3 [1 to 4] | 3 [2.2 to 4]
Statistical Analysis 1: Comparison: Symbiotic vs Distilled Water; Test type: Superiority or Other; p = 0.66, Mann whitney U

4. Primary Outcome: Interleukin 10 Levels at 0+2 Days
Time Frame: 0+2 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 13 [5.5 to 40.5] | 10 [7 to 24]
Statistical Analysis 1: Comparison: Symbiotic vs Distilled Water; Test type: Superiority or Other; p = 0.76, Mann whitney U

5. Primary Outcome: Interleukin 10 Levels at 14+/- 2 Days
Time Frame: 14+/- 2 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 12 [7.5 to 33] | 16 [8 to 28]

6. Primary Outcome: Interleukin 10 Levels at 28+/-2 Days
Time Frame: 28+/-2 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 10 [6 to 13] | 11 [6 to 16]

7. Primary Outcome: Interleukin 17A Levels at 0+2 Days
Time Frame: 0+2 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 1 [1 to 2] | 1 [1 to 1]

8. Primary Outcome: Interleukin 17A Levels at 14+/- 2 Days
Time Frame: 14+/- 2 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 1 [1 to 1.5] | 1 [1 to 2]

9. Primary Outcome: Interleukin 17A Levels at 28+/-2 Days
Time Frame: 28+/-2 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 1 [1 to 1] | 1 [1 to 1.7]

10. Primary Outcome: Interferon Levels at 0+2 Days
Time Frame: 0+2 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 6 [5 to 9.5] | 6.5 [5 to 9.5]

11. Primary Outcome: Interferon Levels at 14+/-2 Days
Time Frame: 14+/-2 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 8 [6 to 11] | 7.5 [7 to 9]

12. Primary Outcome: Interferon Levels at 28+/-2 Days
Time Frame: 28+/-2 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Symbiotic | Distilled Water
Number analyzed (Participants) | 25 | 28
pg/ml | 9 [7 to 12] | 7 [6 to 7.7]

ADVERSE EVENTS:
Time Frame: during trial (0-3 months)
Arm/Group | Symbiotic | Distilled Water
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/28
Other Adverse Events (participants affected / at risk) | 0/25 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No